CLINICAL TRIAL: NCT07174336
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY4064809 Combined With a CDK4/6 Inhibitor and Endocrine Therapy in Adults With HR+, HER2-Advanced Breast Cancer With a PIK3CA Mutation Who Received No Prior Treatment for Advanced Breast Cancer (PIKALO-2)
Brief Title: A Study of Tersolisib (LY4064809/STX-478) With Other Anti-Cancer Treatments in Participants With Advanced Breast Cancer With a Genetic Change (PIK3CA)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27726; J6M-MC-JSGD (Other: Eli Lilly and Company); 2025-522791-92-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: STX-478; PI3K
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — STX-478; ribociclib; palbociclib; abemaciclib; Anastrozole; Letrozole; exemestane; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY4064809 + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 1) (Experimental): LY4064809 given orally in one of two doses in combination with investigator's choice of CDK4/6 inhibitor given orally and ET given orally or intramuscularly
  Interventions: Drug: LY4064809; Drug: Ribociclib; Drug: Palbociclib; Drug: Abemaciclib; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant
- LY4064809 + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 2) (Experimental): LY4064809 given orally in combination with CDK4/6 inhibitor given orally and ET given orally or intramuscularly
  Interventions: Drug: LY4064809; Drug: Palbociclib; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant
- Placebo + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 2) (Placebo Comparator): Placebo given orally in combination with CDK4/6 inhibitor given orally and ET given orally or intramuscularly
  Interventions: Drug: Placebo; Drug: Palbociclib; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: LY4064809 — Administered orally
  Other Names: STX-478; Tersolisib
  Arms: LY4064809 + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 1); LY4064809 + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 2)
Drug: Placebo — Administered orally
  Arms: Placebo + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 2)
Drug: Ribociclib — Administered orally
  Arms: LY4064809 + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 1)
Drug: Palbociclib — Administered orally
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: LY4064809 + CDK4/6 Inhibitor + Endocrine Therapy (ET) (Part 1)
Drug: Anastrozole — Administered orally
Drug: Letrozole — Administered orally
Drug: Exemestane — Administered orally
Drug: Fulvestrant — Administered intramuscular

SUMMARY:
The purpose of the study is to assess the efficacy and safety of the addition of Tersolisib (LY4064809/STX-478) to other anti-cancer drugs as first treatment for advanced hormone receptor-positive (HR+)/human epidermal growth factor receptor 2-negative (HER2-) breast cancer. Participants can remain in the study as long as the drug is helping the cancer without unbearable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Are willing to follow contraception requirements. Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* If assigned female at birth, pre-/peri- and postmenopausal status is allowed. Those with pre- or peri-menopausal status at study entry must agree to use ovarian function suppression with any locally approved gonadotropin-releasing hormone (GnRH) agonist.
* If assigned male at birth with an estrogen receptor positive (ER+) breast cancer diagnosis, they must agree to use hormone suppression with a GnRH agonist.
* Have histologically or cytologically confirmed breast cancer, defined as individuals with

  * locally advanced breast cancer not amenable to curative therapy (for example, surgery) or metastatic disease, and
  * hormone receptors (HR)+/human epidermal growth factor receptor 2 (HER2)- or HR+/HER low defined by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines

    * HR status: Documented ER+ and/or progesterone receptor-positive (PR+) tumor according to ASCO/CAP Guidelines, defined as greater than or equal to (≥)1 percent (%) of tumor cells stained positive based on the most recent tumor biopsy and assessed locally
    * HER status: immunohistochemistry score of 1+ or score of 2+ with a negative Fluorescence In Situ Hybridization (FISH) based on local results as defined in the ASCO/CAP Guidelines
* Have evidence of an activating PIK3CA mutation, detected in tumor or blood samples using an appropriate assay.
* Have measurable disease or non-measurable, evaluable bone disease
* Part 1:

  * Received 0-2 prior systemic treatments for advanced breast cancer not amenable to curative therapy (for example, surgery) or metastatic disease.
  * Up to 1 of these prior systemic treatments may contain chemotherapy
* Part 2:

  * Received 0 prior systemic treatment for advanced breast cancer not amenable to curative therapy (for example, surgery) or metastatic disease.
  * Individuals who are eligible are either

    * Population 1 (P1): Endocrine sensitive

      * newly diagnosed with advanced breast cancer (de novo)
      * relapsed with documented evidence of progression greater than (>)12 months from completion of (neo)adjuvant ET ± cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitor, or
    * Population 2 (P2): Endocrine resistant

      * relapsed with documented evidence of progression less than or equal to (≤)12 months of completing (neo)adjuvant ET ± CDK4/6 inhibitor.
      * if a CDK4/6 inhibitor was included as part of neoadjuvant or adjuvant therapy, progression event must be >12 months since completion of CDK4/6 inhibitor portion of neoadjuvant or adjuvant therapy.

Exclusion Criteria:

* Have an established diagnosis of Type 1 diabetes mellitus or Type 2 diabetes mellitus with hemoglobin A1c (HbA1c) ≥8%, fasting blood glucose (FBG) ≥140 milligrams per deciliter (mg/dL) (7.7 millimoles per liter [mmol/L]), or requiring insulin.
* Have inflammatory or metaplastic breast cancer.
* History of leptomeningeal disease or carcinomatous meningitis.
* Have known and untreated or active central nervous system (CNS) metastases. Exception: Asymptomatic brain or spinal metastases if treated by surgery, surgery plus radiotherapy, or radiotherapy alone with no evidence of radiographic progression or hemorrhage within at least 28 days before randomization and no requirement for anticonvulsants or systemic corticosteroids for at least 28 days before randomization.
* Have received treatment with any local or systemic antineoplastic therapy or investigational anticancer agent within 14 days or 4 half-lives, whichever is longer, prior to randomization up to a maximum washout period of 28 days.
* Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dose more than 10 milligrams [mg] daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization.
* Are pregnant, breastfeeding, or intend to become pregnant during the study or within 6 months of the last dose of study intervention and at least 2 years after the last dose of fulvestrant and/or CDK4/6 inhibitor after the final administration of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
(Part 1): Overall Response Rate (ORR): Percentage of Participants with Confirmed Complete Response (CR) or Partial Response (PR) | Baseline through disease progression or death (Estimated up to 5 years)
  As determined by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1
(Part 2): Progression-Free Survival | Baseline to objective progression or death due to any cause (Estimated up to 5 years)
  Investigator-assessed

SECONDARY OUTCOMES:
(Part 1): Disease Control Rate (DCR) | Baseline through measured progressive disease (Estimated up to 5 years)
  per RECIST v1.1
(Part 1): Time to Response (TTR) | Baseline until the date that measurement criteria for CR or PR (whichever is first recorded) are first met (Estimated as approximately 5 years)
  per RECIST v1.1
(Parts 1 and 2): Duration of Response (DOR) | Date of CR or PR to date of objective disease progression or death due to any cause (Estimated up to 5 years)
  per RECIST v1.1
(Part 1): PFS | Baseline to objective progression or death due to any cause (Estimated up to 5 years)
  per RECIST v1.1
(Parts 1 and 2): Overall Survival (OS) | Baseline to deaths from any cause (Estimated up to 7 years)
(Part 1): Best Overall Response (BOR) | Baseline to disease progression or death from any cause (Estimated up to 5 years)
(Parts 1 and 2): Clinical Benefit Rate (CBR): Percentage of Participants with a BOR of CR or PR, or SD Lasting Greater than or Equal to Six Months | Baseline to disease progression or death from any cause (Estimated up to 5 years)
  per RECIST v1.1
(Parts 1 and 2): PK: Average Plasma Concentrations of LY4064809 | Baseline to last PK sample collection up to 5 months
(Part 2): Progression-Free Survival after Subsequent Line of Treatment (PFS2) | Baseline to disease progression on next line of treatment or death from any cause (Estimated as up to 7 years)
  Investigator-assessed
(Part 2): Progression-Free Survival (PFS) | Baseline to objective progression or death from any cause (Estimated up to 5 years)
  By BICR
(Part 2): Objective Response Rate (ORR) | Baseline to disease progression or death from any cause (Estimated up to 5 years)
  By investigator and blinded independent central review (BICR)
(Part 2): Time to Chemotherapy (TTC) | Baseline until the start of chemotherapy (Estimated up to 7 years)
(Part 2): Chemotherapy-Free Survival | Baseline until the start of chemotherapy or death from any cause (Estimated up to 7 years)
(Part 2): Change in Overall Health-related Quality of Life (HRQoL) as measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status/Quality of Life Subscale | Baseline until disease progression or death (Estimated up to 7 years)
  The EORTC QLQ-C30 is a 30-question patient-reported instrument used to assess multidimensional HRQoL in cancer patients. Overall HRQoL is measured by the EORTC QLQ-C30 Global Health Status/Quality of Life Subscale (two items). Response options range from 1) "very poor" to 7) "excellent." Score is linearly transformed to the range 0 - 100. Higher score represents better overall HRQoL.
(Part 2): Change in Physical Function as measured by the EORTC QLQ-C30 Physical Functioning Subscale | Baseline until disease progression or death (Estimated up to 7 years)
  The EORTC QLQ-C30 is a 30-question patient-reported instrument used to assess multidimensional HRQoL in cancer patients. Physical function is measured by the EORTC QLQ-C30 Physical Functioning subscale (five items). Response options range from 1) "not at all" to 4) "very much." Score is linearly transformed to the range 0 - 100. Higher score represents better overall physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (276):
- United States (86):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Marin Cancer Care, Greenbrae, California
  - Chao Family Comprehensive Cancer Center and Ambulatory Care (CIACC) - Irvine, Irvine, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente Oakland, Oakland, California
  - Profound Research LLC, Oceanside, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Center, Palo Alto, California
  - Kaiser Permanente, Roseville, California
  - Kaiser Permanente, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Kaiser Permanente, Santa Clara, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Kaiser Permanente, Vallejo, California
  - Kaiser Permanente Walnut Creek, Walnut Creek, California
  - Clermont Oncology Center, Clermont, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Summit Cancer Care, PC, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Accellacare of Duly, Lisle, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Saint Elizabeth Medical Center Edgewood, Edgewood, Kentucky
  - Our Lady of the Lake RMC, Baton Rouge, Louisiana
  - American Oncology Partners, PA, Bethesda, Maryland
  - James M Stockman Cancer Institute, Frederick, Maryland
  - Mass General Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center - South Shore Hospital, South Weymouth, Massachusetts
  - Profound Research LLC, Sterling Heights, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - North Mississippi Hematology and Oncology Associates, Tupelo, Mississippi
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Jefferson Health - Cherry Hill, Cherry Hill, New Jersey
  - Sidney Kimmel Cancer Center - Washington Township, Sewell, New Jersey
  - Atlantic Health System Overlook Medical Center, Summit, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - WakeMed Cancer Care - Waverly Hematology & Medical Oncology, Cary, North Carolina
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Carolina Cancer Research Center, Wilson, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer -T, Columbus, Ohio
  - Cleveland Clinic - Hillcrest Hospital, Mayfield Heights, Ohio
  - Good Samaritan Regional Medical Center, Corvallis, Oregon
  - Oncology Associates of Oregon, Eugene, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Jefferson Hospital Northeast, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Nashville General Hospital, Nashville, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - World Research Link, Baytown, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - USO - Texas Oncology, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - West Texas, El Paso, Texas
  - Oncology Consultants P.A., Houston, Texas
  - Nova Oncology, McAllen, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - US Oncology Research Network, The Woodlands, Texas
  - Tranquility Research, Webster, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Swedish Cancer Institute - Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - UW Medicine Valley Medical Center, Renton, Washington
  - Swedish Medical Center, Seattle, Washington
  - Cancer Care Northwest - Vercler, Spokane Valley, Washington
  - ThedaCare Physicians - Appleton North, Appleton, Wisconsin
- Argentina (10):
  - CIPREC, Buenos Aires
  - Investigaciones Clinicas Moleculares (ICM), Buenos Aires
  - Centro Oncologico Korben, Buenos Aires
  - Hospital Medico Policial Churruca-Visca, Buenos Aires
  - Organizacion Medica de Investigacion, Buenos Aires
  - Fundación Innovaciencia, Rosario
  - Hospital Provincial del Centenario, Rosario
  - COE (Centro Oncológico de Excelencia), San Juan
  - Instituto San Marcos, San Juan
  - Go Centro Medico San Nicolás, San Nicolás
- Australia (8):
  - The Prince Charles Hospital, Brisbane
  - St Vincent's Hospital, Darlinghurst
  - Peter MacCallum Cancer Centre, Melbourne
  - Lake Macquarie Private Hospital, Newcastle
  - Macquarie University, North Ryde
  - Goulburn Valley Health, Shepparton
  - St. John of God Subiaco Hospital, Subiaco
  - The Townsville Hospital, Townsville
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - AZ Nikolaas, Sint-Niklaas
- Brazil (15):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Hospital São Domingos, Bequimão
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará, Fortaleza
  - Hospital Araújo Jorge, Goiânia
  - Hospital Brasilia, Lago Sul
  - Hospital de Cancer de Londrina, Londrina
  - Instituto Atena de Pesquisa Clinica - Mossoró, Mossoró
  - Liga Norte Riograndense Contra o Câncer, Natal
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Centro de Tratamento de Tumores Botafogo para Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital Santa Catarina - Paulista, São Paulo
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
- Canada (3):
  - Hamilton Health Sciences-Juravinski Cancer Centre, Hamilton
  - CHU de Québec-Université Laval, Hôpital du Saint-Sacrement, Québec
  - Princess Margaret Cancer Centre, Toronto
- China (21):
  - Anyang Cancer Hospital, Anyang
  - Beijing Cancer hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - Deyang City People's Hospital, Deyang
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangmen Center Hospital, Jiangmen
  - The first affiliated hospital of Ningbo university, Ningbo
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
  - Central Hospital of Guangdong Provincial Agricutural Reclamation, Zhanjiang
- France (13):
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - CHU Besançon, Besançon
  - CHRU de Brest, Brest
  - Clinique Victor Hugo Le Mans, Le Mans
  - Hopital Prive Jean Mermoz, Lyon
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Institut Curie - site Saint-Cloud, Saint-Cloud
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Oncopole Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (23):
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Marienhospital Bottrop, Bottrop
  - Universitaetsklinikum Koeln, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Onkologiezentrum Donauwörth, Donauwörth
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - MVZ Medical Center Düsseldorf GmbH, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Private Practice - Dr. Helmut Oettle und Prof.Dr.med. Frank Mayer, Friedrichshafen
  - OSP Göttingen, Göttingen
  - Mammazentrum HH - Krankenhaus Jerusalem, Hamburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
  - Klinikum Ernst von Bergmann, Potsdam
  - Helios HSK Wiesbaden, Wiesbaden
  - Marien Hospital Witten, Witten
  - HELIOS Klinikum Wuppertal, Wuppertal
- Greece (8):
  - Agios Savvas Regional Cancer Hospital, Athens
  - Aretaieio Hospital, Athens
  - Attikon General University Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - European Interbalkan Medical Center, Thessaloniki
- Italy (12):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Humanitas Istituto Clinico Catanese, Misterbianco
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Japan (14):
  - Kyushu University Hospital, Fukuoka
  - Hiroshima City Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Sagara Hospital, Kagoshima
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Kyoto University Hospital, Kyoto
  - Kanazawa Medical University Hospital, Mukai-awagasaki
  - Nagoya City University Hospital, Nagoya
  - Nakagami Hospital, Okinawa
  - Gunma Prefectural Cancer Center, Otashi
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Showa Medical University Hospital, Shinagawa City
  - Tsukuba University Hospital, Tsukuba
- South Korea (10):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si
  - Kyungpook National University Chilgok Hospital, Deagu
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu
  - Yeungnam Univeristy Medical Center, Gyeongsan-si
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (26):
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario San Cecilio, Granada
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Beata María Ana, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (8):
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Adana City Hospital, Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Ege Universitesi Hastanesi, Bornova
  - Trakya University, Edirne
  - Koç Üniversitesi Hastanesi, Istanbul
  - Yeditepe Üniversitesi Koşuyolu Hastanesi, Istanbul
- United Kingdom (7):
  - Huddersfield Royal Infirmary, Huddersfield
  - St Bartholomew's Hospital, London
  - Royal Marsden Hospital (Sutton), London
  - Royal Marsden Hospital (Chelsea), London
  - The Christie NHS Foundation Trust, Manchester
  - Derriford Hospital, Plymouth
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/